CLINICAL TRIAL: NCT07223710
Title: Engaging Reticulospinal Inputs to Improve Walking Ability in Humans With Spinal Cord Injury
Brief Title: Improving Walking After Spinal Cord Injury
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dalia DeSantis, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00222004; R03HD114768-01 (NIH)
Record Dates: First submitted 2025-10-27; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury
Keywords: auditory stimulation; peripheral stimulation; locomotion training; descending motor tracts
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locomotor training + PAS (Experimental): This intervention uses repeated paired loud auditory and electrical stimulation of muscle afferents combined with locomotor training.
  Participants will exercise walking on a treadmill with body weight support as needed for 30 minutes a day at a moderate intensity. While walking, participants will receive brief loud auditory stimuli through headphones and short electrical pulses through of electrodes positioned on two points in the leg
  Interventions: Device: Paired Associative Stimulation; Behavioral: Locomotor Training
- Locomotor training + SHAM (Sham Comparator): This sham intervention uses repeated paired soft auditory clicks and electrical stimulation of muscle afferents combined with locomotor training.
  Participants will exercise walking on a treadmill with body weight support as needed for 30 minutes a day at a moderate intensity. While walking, participants will receive brief auditory clicks through headphones and short electrical pulses through a pair of electrodes positioned on two points in the leg.
  Interventions: Behavioral: Locomotor Training; Device: Sham stimulation

INTERVENTIONS:
Device: Paired Associative Stimulation — This new intervention consists of locomotor training in combination with paired low-intensity electrical stimulation and stimulation of the reticulospinal tract through loud sounds. Participants will receive auditory stimulation (LAS, 110dB, 500Hz, 50ms) through headphones and electrical stimulation through a pair of electrodes with 2cm inter-electrode distance positioned on the motor point over the quadriceps and the tibialis anterior muscles bilaterally. The motor point will be identified as the position of the electrodes that elicits a small visible muscle twitch or muscle contraction upon palpation over the tendon with the minimum stimulation intensity. Stimuli will be delivered with a pulse duration of 200 microseconds and will be timed to arrive at the level of the brainstem ~7ms before auditory signals.
  Other Names: PAS
  Arms: Locomotor training + PAS
Behavioral: Locomotor Training — Participants will walk on a treadmill with body-weight support (ZeroG, Aretech) in the range 0-70% as needed to prevent excessive knee flexion during stance phase or toe dragging during swing phase (Finch et al. 1991). Each session will last approximately 60-min and the duration of the treadmill training will be timed to be 30 min. Subjects will be encouraged to walk at a self-selected speed at or above 0.1m/s. Speed and body-weight support will be adjusted to achieve a perceived exertion score of 4-5 (Moderate) in the Borg scale (Borg 1982). Subjects will be allowed to rest as needed during the training sessions.
Device: Sham stimulation — Participants will receive brief low-intensity auditory clicks (80dB, 500Hz, 50ms) through headphones and electrical stimulation through a pair of electrodes with 2cm inter-electrode distance positioned on the motor point over the quadriceps and the tibialis anterior muscles bilaterally. The motor point will be identified as the position of the electrodes that elicits a small visible muscle twitch or muscle contraction upon palpation over the tendon with the minimum stimulation intensity. Stimuli will be delivered with a pulse duration of 200 microseconds and will be timed to arrive at the level of the brainstem ~7ms before auditory signals.
  Arms: Locomotor training + SHAM

SUMMARY:
Locomotor recovery is one of the most important goals of individuals with spinal cord injury (SCI). Ambulatory deficits severely impact daily functions resulting in lower quality of life for people living with paralysis due to SCI. Although studies have shown that locomotor training improves locomotor function in people with chronic SCI, the benefits remain limited. Our overall hypothesis is that we can engage additional descending motor pathways, such as the reticulospinal tract (RST), to improve locomotor function in humans with chronic incomplete SCI.

In this study we propose to test the effects of a novel intervention that uses repeated paired loud auditory and electrical stimulation of muscle afferents combined with locomotor training on walking speed and voluntary muscle strength.

DETAILED DESCRIPTION:
Individuals with chronic incomplete SCI will be randomly assigned to a group that will receive 10 sessions of a startle stimulus (a very brief, loud sound) and electrical stimulation combined with locomotor training or 10 sessions of a non-startle stimulus (a very brief, soft sound) combined with locomotor training.

ELIGIBILITY:
Inclusion Criteria:

* History of traumatic or non-traumatic SCI ≥ 6 months
* International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) level at and above T10.
* American Spinal Injury Association AIS Grade C, or D
* Weakness in ankle dorsiflexors (LEMS<=3) with the ability to perform a small voluntary ankle dorsiflexion (as detected by presence of voluntary EMG activity in the tibialis anterior) with at least one leg.
* Ability to tolerate standing position.
* Ability to walk at a minimum speed of 0.1 mile/hour on a treadmill with less than 70% body weight support.
* Requires use of assistive devices (KAFO, AFO, cane, walker) or body weight support for ambulation.
* Ability to complete the 10-Meter Walk Test.

Exclusion Criteria:

* Preceding uncontrolled medical conditions including pulmonary, cardiovascular or orthopedic disease that interfere with physical performance.
* Intolerance to physical activity.
* Severe cognitive impairment that precludes the ability to participate in any of the study procedures or give verbal consent.
* Any illness or condition that based on the research team's assessment, will compromise with the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during the study.
* History of stroke resulting in sensory motor deficits.
* Pregnant women.
* Participation in a high-intensity locomotor training program in the last 6 months.
* Inability to detect somatosensory evoked potentials
* Metal implant in the head
* History of epilepsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
10-meter walk test (10MWT) | baseline and day 12
  This standardized test assesses walking speed in meters per second over a short duration.

SECONDARY OUTCOMES:
Motor Evoked Potentials conditioned with Startle (MEP-LAS) | Baseline and day 12
  Motor Evoked Potentials (MEPs) will be recorded from multiple leg muscles following transcranial magnetic stimulation over the leg representation of the primary motor cortex and electrical stimulation over the thoracic spine. Loud auditory Stimuli (LAS, 110dB, 500Hz, 50ms) will be delivered 50ms before magnetic stimulation to test for cortical effects of the intervention and 80ms before the electrical stimulation to test for subcortical effects of the intervention. Stimulation intensity will be adjusted to obtain unconditioned MEPs of ~50% of the maximum MEP for each muscle.
Maximum Voluntary Contraction (MVC) | Baseline and day 12
  This will be measured on the electromyographic signal recorded during maximal isometric contractions. Participants will perform three maximal contractions against resistance into knee flexion and extension, dorsiflexion, and plantarflexion. Electromyographic activity will be monitored using surface electrodes placed on the belly of the quadriceps femoris, hamstrings, tibialis anterior, and soleus muscles bilaterally. The MVC will be quantified as the maximum value of the average over 1s of activity in each of the repetitions.
Maximal motor response (M-max) | Baseline and day 12
  M-max will be elicited in the quadriceps femoris, tibialis anterior, soleus and foot muscles by applying percutaneous electrical stimulation over the femoral, common peroneal and the tibial and the medial plantar nerve, respectively using 200μs rectangular electrical stimulus. The intensity of stimulation will be increased progressively until M-max is reached.
StartReact response | Baseline and day 12
  Participants will be asked to observe a light-emitting diode (LED) located ~1 m in front of the participants' head and will be wearing headphones. When the LED will illuminate (20 ms), individuals will be asked to perform an isometric knee flexion/extension and/or ankle dorsi/plantarflexion as fast as possible. Reaction times will be evaluated following a visual cue either alone (20 trials) or paired with a non-startling (80dB, 500Hz, 50ms, 20 trials) or a startling (110dB, 500Hz, 50ms, 20 trials) auditory cue. Stimuli will be delivered every 5s in a randomized order. Target muscles will be quadriceps femoris, hamstrings, tibialis anterior, and soleus muscles of the weaker leg. The StartReact response will be computed as the difference between the reaction times during a non-startling and startling auditory cue
Spasticity | Baseline and day 12
  We will use the Modified Ashworth scale (six-point ordinal scale, 0-4) to measure resistance encountered during manual passive muscle stretching.
SCI-QOL | Baseline and day 12
  Is a battery of questionnaires evaluating the quality of life. Will be used to measure the participant-related following aspects: (a) Ambulation: This questionnaire will ask the participant about their ability to do thing like walk, run and jump. (b) Basic Mobility: This questionnaire will ask the participant about their ability to perform their daily routine. (c) Fine Motor: This questionnaire will ask the participant about their ability to pick up small objects. (d) Manual and Power Wheelchair Mobility: This questionnaire ask the participant about their ability using a wheelchair. (e) Self-Care: This questionnaire will ask the participant about their ability to do activities of daily living such as getting dressed, bathing, and eating.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia De Santis, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to Demographics, clinical outcomes and instrumental data will shared through the NICHD Data ad Specimens Hub (DASH).
Supporting Information: Study Protocol
Time Frame: The de-identified IPD will be shared indefinitely on DASH. The data will be available at the end of the study.